CLINICAL TRIAL: NCT00378417
Title: Efficacy Trial in Finnish Children of Two Pneumococcal Conjugate Vaccines (PncCRM and PncOMPC) for Prevention of Acute Otitis Media Due to Pneumococcal Serotypes in the Vaccines
Brief Title: Efficacy Trial of Two Pneumococcal Conjugate Vaccines (PncCRM and PncOMPC) for Prevention of Acute Otitis Media Due to Vaccine Serotypes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Wyeth-Lederle Vaccines (Industry); Pasteur Merieux Connaught (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KTL69-0; PNC95KTL
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Otitis Media; Pneumococcal Infections
Keywords: Otitis Media; Pneumococcal Infections; Pneumococcal Vaccines; Proportional Hazards Models; Prospective Studies; Streptococcus pneumoniae; Vaccines, Conjugate
MeSH Terms: conditions — Otitis Media; Pneumococcal Infections

INTERVENTIONS:
Biological: 7-valent pneumococcal-CRM197 conjugate vaccine
Biological: 7-valent pneumococcal-OMPC conjugate vaccine

SUMMARY:
This was a randomized, double-blinded multicenter cohort study of Finnish children aged 2 to 24 months. The study was designed to evaluate the efficacy of two 7-valent pneumococcal conjugate vaccines (PncCRM and PncOMPC) parallelly, both vaccines compared with the same control vaccine (hepatitis B vaccine).

The primary endpoint was culture-confirmed pneumococcal acute otitis media (AOM) episodes due to all serotypes included in the pneumococcal conjugate vaccine and the primary hypothesis was that, compared to the control vaccine group, the pneumococcal conjugate vaccine would protect infants from culture confirmed AOM caused by pneumococcal serotypes in the vaccine. The efficacy of the two vaccines against any pneumococcal AOM and any AOM was also evaluated.

The children were vaccinated with the pneumococcal conjugate vaccine or the control vaccine at the age of 2, 4, 6 and 12 months and followed at study clinics established specifically for the purpose from 2 to 24 months of age. Whenever AOM was diagnosed during the follow-up, middle ear fluid was aspirated for bacterial culture.

ELIGIBILITY:
Inclusion Criteria:

* infants coming to their own child health center before the age of 13 weeks, and judged to be in good health on the basis of medical history and physical examination
* family living permanently in Tampere, Kangasala or Nokia
* at least one of the parents/guardians is able to communicate fluently in Finnish
* written informed consent obtained from a parent/guardian prior to enrollment in the study

Exclusion Criteria:

* hypersensitivity to any of the components of the vaccines used in the study,
* known or suspected impairment of immunologic function,
* history of invasive pneumococcal disease,
* prior vaccination with any pneumococcal vaccine,
* prior vaccination with hepatitis B vaccine,
* contraindications to routine childhood immunizations
* any medical condition in which, in the opinion of the investigator, the study procedures or vaccinations might cause risk to the health or endanger the well-being of the child

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3075
Dates: Start 1995-03; Study Completion 1999-03

PRIMARY OUTCOMES:
Culture-confirmed pneumococcal acute otitis media episodes due to all serotypes included in the pneumococcal conjugate vaccine

SECONDARY OUTCOMES:
First episodes of culture-confirmed pneumococcal AOM due to all serotypes included in the pneumococcal conjugate vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Eskola, MD, Principal Investigator — Finnish Institute for Health and Welfare; Terhi Kilpi, MD, Study Director — Finnish Institute for Health and Welfare
Locations (5):
- Finland (5):
  - Kangasala Study Clinic, Kangasala
  - Nokia Study Clinic, Nokia
  - Eteläinen, Keskinen, and Läntinen Study Clinic, Tampere
  - Itäinen and Pohjoinen Study Clinic, Tampere
  - Kaakkoinen Study Clinic, Tampere

REFERENCES:
- [Result] Eskola J, Kilpi T, Palmu A, Jokinen J, Haapakoski J, Herva E, Takala A, Kayhty H, Karma P, Kohberger R, Siber G, Makela PH; Finnish Otitis Media Study Group. Efficacy of a pneumococcal conjugate vaccine against acute otitis media. N Engl J Med. 2001 Feb 8;344(6):403-9. doi: 10.1056/NEJM200102083440602. PMID 11172176
- [Result] Kilpi T, Ahman H, Jokinen J, Lankinen KS, Palmu A, Savolainen H, Gronholm M, Leinonen M, Hovi T, Eskola J, Kayhty H, Bohidar N, Sadoff JC, Makela PH; Finnish Otitis Media Study Group. Protective efficacy of a second pneumococcal conjugate vaccine against pneumococcal acute otitis media in infants and children: randomized, controlled trial of a 7-valent pneumococcal polysaccharide-meningococcal outer membrane protein complex conjugate vaccine in 1666 children. Clin Infect Dis. 2003 Nov 1;37(9):1155-64. doi: 10.1086/378744. Epub 2003 Oct 7. PMID 14557958
- [Derived] Ekstrom N, Ahman H, Palmu A, Gronholm S, Kilpi T, Kayhty H; FinOM Study Group. Concentration and high avidity of pneumococcal antibodies persist at least 4 years after immunization with pneumococcal conjugate vaccine in infancy. Clin Vaccine Immunol. 2013 Jul;20(7):1034-40. doi: 10.1128/CVI.00039-13. Epub 2013 May 8. PMID 23658394